CLINICAL TRIAL: NCT06914141
Title: Comparative Effectiveness of Tirzepatide Versus Semaglutide in Individuals With Heart Failure With Preserved Ejection Fraction
Acronym: DUP-TIRZSEMA
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TIRZSEMA
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; HFpEF - Heart Failure With Preserved Ejection Fraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tirzepatide: New use of tirzepatide dispensing claim is used as the exposure.
  Interventions: Drug: Tirzepatide
- Semaglutide: New use of semaglutide dispensing claim is used as the reference.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — New use of tirzepatide dispensing claim is used as the exposure.
  Groups: Tirzepatide
Drug: Semaglutide — New use of semaglutide dispensing claim is used as the reference.
  Groups: Semaglutide

SUMMARY:
Investigators are building an empirical evidence base for real-world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of tirzepatide vs semaglutide after emulating the pivotal RCTs of each drug used to support regulatory approval in heart failure with preserved ejection fraction (SUMMIT and STEP-HFpEF DM trials).This comparative effectiveness target trial described below draws from eligibility criteria from the SUMMIT and STEP-HFpEF DM trials. Although many features of the target trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The database study will be a new-user active-comparative study, conducted using 2 national United States claims databases, where we compare the effect of tirzepatide vs semaglutide on the composite end point of all-cause mortality or heart failure hospitalization. Clinical guidelines during the study period recommended both agents for the same indications of glucose lowering and weight reduction. Indication for heart failure with preserved ejection fraction has not been granted for both drugs during the study period.

ELIGIBILITY:
Eligible cohort entry dates:

Optum: Study period between May 13, 2022 to November 30, 2024. Marketscan: Study period between May 13, 2022 to December 31, 2023.

Inclusion Criteria:

* Heart failure
* BMI > 27.0 kg/m2
* History of type 2 diabetes mellitus
* LVEF ≥ 45%
* ≥ 18 years old, male or female sex

Exclusion Criteria:

* Prior treatment with any GLP-1-RA
* History of type 1 diabetes mellitus
* End-stage renal disease or chronic or intermittent haemodialysis or peritoneal dialysis
* History of bariatric surgery
* History of nursing home admission
* Pregnant female or breastfeeding
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy
* Treatment with continuous subcutaneous insulin infusion
* Multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinoma of the cervix, or in situ prostate cancer) for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals aged 40 years or older with heart failure with preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 28118 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality or heart failure hospitalization | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on all-cause mortality or heart failure hospitalization in patients with heart failure with preserved ejection fraction.

SECONDARY OUTCOMES:
Composite of all-cause mortality or all-cause mortality or a worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization, intravenous diuretic therapy in an urgent care setting). | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on all-cause mortality or worsening heart failure events in patients with heart failure with preserved ejection fraction.
Worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting). | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on worsening heart failure event (exacerbated symptoms of heart failure resulting in hospitalization or intravenous diuretic therapy in an urgent care setting) in patients with heart failure with preserved ejection fraction.
Intravenous diuretic therapy in an urgent care setting | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on intravenous diuretic therapy in an urgent care setting in patients with heart failure with preserved ejection fraction.
Hospitalization for heart failure | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on hospitalization for heart failure in patients with heart failure with preserved ejection fraction.
All-cause mortality | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on all-cause mortality in patients with heart failure with preserved ejection fraction.
Urinary tract infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on urinary tract infection in patients with heart failure with preserved ejection fraction.
Serious bacterial infection | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on serious bacterial infection in patients with heart failure with preserved ejection fraction.
Gastrointestinal adverse events | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the comparative effect of tirzepatide vs semaglutide on gastrointestinal adverse events in patients with heart failure with preserved ejection fraction.

OTHER OUTCOMES:
Hernia | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs semaglutide on a negative control outcome of hernia.
Lumbar radiculopathy | Through study completion (1 day after cohort entry date until the first of outcome or censoring)
  To evaluate the effect of tirzepatide vs semaglutide on a negative control outcome of lumbar radiculopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Fuse K, Matseyko S, Sreedhara SK, Hahn G, Schunkert H, Wang SV. Semaglutide and Tirzepatide in Patients With Heart Failure With Preserved Ejection Fraction. JAMA. 2025 Oct 14;334(14):1255-1266. doi: 10.1001/jama.2025.14092. PMID 40886075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT06914141/Prot_SAP_000.pdf